CLINICAL TRIAL: NCT05981638
Title: Investigation of the Effect of Mobilization on Gastric Emptying Time Among Pediatric Patients Scheduled for Elective Surgery: Randomised Controlled Trial
Brief Title: The Effect of Mobilization on Gastric Emptying Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Cansabuncu, principal investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-7/26
Record Dates: First submitted 2023-06-08; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia; Fasting
Keywords: diagnostic imaging; fasting; anesthesia
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group WM (Water+mobilization) (Other): All patients were randomized according to a table created on a computer using the closed-envelope method.Patients in the WM group (water+mobilization) were given water and mobilized
  Interventions: Other: group WM
- Group WR(water+rest) (Other): All patients were randomized according to a table created on a computer using the closed-envelope method. Patients in the WR group (water+rest) were given water and stay in rest
  Interventions: Other: group WR
- Group AR(apple juice+rest) (Other): All patients were randomized according to a table created on a computer using the closed-envelope method. Patients in the AR group (apple juice+rest) were given apple juice and stay in rest
  Interventions: Other: Group AR
- Group AM (apple juice+mobilization) (Other): All patients were randomized according to a table created on a computer using the closed-envelope method. Patients in the AM group (apple juice+mobilization) were given water and mobilized
  Interventions: Other: Group AM

INTERVENTIONS:
Other: group WM — Patients were given 5ml/kg dose of water and patients were mobilized.
  Arms: Group WM (Water+mobilization)
Other: group WR — Patients were given 5ml/kg dose of water and patients were rest.
  Arms: Group WR(water+rest)
Other: Group AR — Patients were given 5ml/kg dose of apple juice and patients were rest.
  Arms: Group AR(apple juice+rest)
Other: Group AM — Patients were given 5ml/kg dose of apple juice and patients were mobilized.
  Arms: Group AM (apple juice+mobilization)

SUMMARY:
ıntroduction Pulmonary aspiration under general anesthesia is a rare but serious complication in healthy patients undergoing elective surgery. In the preoperative period, negative metabolic, physiological, and/or psychological consequences may occur due to prolonged hunger time (1). It is important to shorten the preoperative fasting period to reduce anxiety and hunger, especially in pediatric patients (2).

Material-Methods This study at Bursa Uludag University Hospital (January 2021- January 2022) involved 84 ASA (American Society of Anesthesiologists) class I-III patients aged 4-11 years undergoing elective urogenital surgery, with certain exclusions like gastrointestinal disorders and high BMI (Body Mass Index).

Gastric antral area (GAA) was measured with ultrasound (USG) before liquid intake and at various intervals there after; 5, 10, 30, 60, 90 minutes. Patients were split into four groups based on liquid (water or apple juice) and activity level (rest or mobilization). Resting patients watched animations, while mobilized patients were encouraged to walk.

DETAILED DESCRIPTION:
This prospective study was carried out at Bursa Uludag University Hospital between January 2021 and January 2022, following the approval of the local ethical committee (2021-7/26). Eighty-four ASA class I-III patients aged 4-11 years who were scheduled for elective urogenital surgery were included in the study. The parents were informed about the research, both verbally and in writing, and their consent was obtained. Patients with a pathology that prevents emptying in the upper gastrointestinal system, who have motility disorders in the gastrointestinal system, who are under follow-up due to diabetes mellitus (DM), who can-not cooperate, refuse to drink fluids or USG, do not provide consent from their families, have a history of lower esophagus or gastric operation, have a history of upper gastrointestinal bleeding in the last month, clinically significant hepatic or renal failure, and a BMI > 35 kg m2 were excluded from the study.During the preoperative visit, the child's physical characteristics (sex, age, weight, height, and body mass index) and initial vital parameters (heart rate and noninvasive blood presure) were recorded. Oral intake was discontinued in all children according to our common protocol (two hours for clear liquids; six hours for semi-solid and solid foods)All patients were randomized according to a table created on a computer using the closed-envelope method. It was planned such that only the surgeons knew which group the randomized patients were in. The anesthesiologist who performed the USG measurements did would not know which group the patient belonged to. Informed consent was obtained after the study protocol was properly explained to the children in accordance with their parents and age. In the clinic, clear liquids (water or apple juice) at room temperature (22°C) were administered to the patients by a second anesthesiologist and clinic nurse, in accordance with the group. The gastric antral area (GAA) was measured with USG just before the intake of liquid (T0), at the 5th minute (T5), 10th minute (T10), 30th minute (T30), 60th minute (T60), 90th minute (T90) by the anesthesiologist. This planned procedure was performed on the morning of the day of the operation, at least two hours before the induction of anesthesiaThe patients were grouped according to the kind of liquid (water or apple juice) and physical activity (resting or mobilization). [Group WR [water+rest (n:19)], Group WM [water+mobilization (n:21)], Group AR [apple juice (49.6kcal/100 ml + rest (n:23)] and Group AM [apple juice (49.6kcal/100 ml) + mobilization (n:21)]]. All the clear liquids were administered at a dose of 5 ml/kg. Patients in the resting groups (WR and AR); sat between ultrasound examinations and watched the age-appropriate animation of their choice. Age-appropriate audiovisual interventions such as cartoons and interactive games are effective in reducing preoperative anxiety in children. However, the selection of audiovisual interventions according to the age of the child is crucial. Patients in the mobilized group (WM and AM) were encouraged to walk into the clinic and their rooms between the ultrasound examinations.During USG imaging, patients were placed in a 45° semi-recumbent, right lateral decubitus (RLD) position. A portable ultrasound device (Logic E® GE, Boston, MA, USA) equipped with a high-frequency linear array transducer (probe 8-12 MHz) was used to obtain a cross-sectional image of the gastric antrum. The gastric antrum was identified in the sagittal or sagittal oblique plane in the epigastrium, along the edge of the left lobe of the liver, and anterior to either the aorta or the inferior vena cava, according to the standard protocol. Gastric emptying is influenced by gravity and should be faster in an upright positionGAA, craniocaudal (D1) (cm) and anteroposterior (D2) (cm) of the antrum, including stomach wall, in the RLD position werw calculated using real-time USG (Logic E® GE, Boston, USA) linear probe (8-12 MHz) diameters. A single cross-section of the antrum was obtained in the sagittal plane containing the left lobe of the liver and the aorta or inferior vena cava and was considered a standard level for measuring craniocaudal and anteroposterior diameters. The values of these diameters were inserted into the formula below to calculate the antral GAA, which correlates with gastric volume (GAA = π × D1 × D2/4).

A single investigator evaluated the hunger and thirst ratings of all children before drinking the beverages (0 min), and at 10, 15, 30, 60, and 90 min after drinking.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III patients aged 4-11 years who were scheduled for elective urogenital surgery were included in the study.

Exclusion Criteria:

* Patients with pathology that prevents emptying in the upper gastrointestinal system, who have motility disorders in the gastrointestinal system, who are under follow-up due to diabetes mellitus (DM), who can not cooperate, who refuse to drink fluids or USG, who do not give consent from their families, who have a history of the lower esophagus or gastric operation, with a history of upper gastrointestinal bleeding in the last one month, clinically significant hepatic or renal failure, and a BMI > 35 kg m2 were excluded from the study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Measurement of gastric antral area change with USG within 90 minutes after clear fluid intake | Baseline and after clear fluid intake at 10, 15, 30, 60, and 90 minutes
  Ultrasonography (USG) is a non-invasive and reliable imaging method that can be used to measure stomach content. It is widely used to examine the gastric antral cross-sectional area (GAA) (cm2) in adult and pediatric patients.The purpose of this study was to investigate the effect of mobilization and the type of liquid drink (drinking water or apple juice) on gastric emptying time among pediatric patients scheduled for elective surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Cansabuncu, Principal Investigator — BURSA ULUDAG UNIVERSITY HOSPITAL; Selcan Akesen, Study Chair — BURSA ULUDAG UNIVERSITY HOSPITAL; Belgin Yavaşcaoğlu, Study Chair — BURSA ULUDAG UNIVERSITY HOSPITAL; Fatih Çelik, Study Chair — BURSA ULUDAG UNIVERSITY HOSPITAL
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)